CLINICAL TRIAL: NCT07177599
Title: Global, Regional, and National Burdens of Pancreatic Cancer and Pancreatitis Among Older Adults From 1990 to 2021 With Projections to 2040: A Comprehensive and Comparative Investigation
Brief Title: Pancreatic Disease Burden in Older Adults (1990-2040)
Status: Completed | Type: Observational
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Huang Hai, Prof. Dr., Changhai Hospital
Other Study IDs: GePCPS-01
Record Dates: First submitted 2025-09-10; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Pancreatic Cancer; Pancreatitis
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pancreatic Cancer
  Interventions: Biological: Natural history
- Pancreatitis
  Interventions: Biological: Natural history

INTERVENTIONS:
Biological: Natural history — Natural history of pancreatic diseases

SUMMARY:
Using data from the Global Burden of Disease Study 2021, the investigators analyzed age-standardized incidence, mortality, and disability-adjusted life-years (DALYs) for pancreatic cancer and pancreatitis in adults aged ≥70 years across 204 countries and territories, stratified by sex, Socio-Demographic Index (SDI), health system performance, and region. The investigators calculated estimated annual percentage changes (EAPCs), applied age-period-cohort modelling, and used Bayesian models to project future burden. Attributable burdens for key risk factors were also estimated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis with pancreatic cancer or pancreatitis
* Diagnosis in 1990 through 2021
* Age 70+ years

Exclusion Criteria:

* Age <70 years
* Other non-pancreatic diseases

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study population consisted of patients aged 70 years or older who were diagnosed with either pancreatic cancer or pancreatitis between 1990 and 2021. Individuals under the age of 70 were excluded from participation. Additionally, those with comorbid non-pancreatic diseases were also excluded to minimize potential confounding effects and to maintain a focus on conditions specifically related to the pancreas.
Sampling Method: Probability Sample
Enrollment: 723415 (Actual)
Dates: Start 1990-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2025-09-11 (Actual)

PRIMARY OUTCOMES:
Incidence | 1990-2021
  The number of new cases of a givencause during a given period in aspecified population. It is xpressed as the number of newcases in a year divided by the mid-year population size.
Deaths | 1990-2021
  Deaths occurring in a population during a certain time period.
Disability-adjusted life years (DALYs) | 1990-2021
  The sum of years lost due to premature death (YLLs) and yearslived with disability (YLDs). DALYs are also defined as years of healthy life lost.